CLINICAL TRIAL: NCT00327730
Title: Evaluation of Eperisone HCl in the Treatment of Acute Musculoskeletal Spasm Associated With Low Back Pain
Brief Title: Evaluation of Eperisone HCl in the Treatment of Acute Musculoskeletal Spasm Associated With Low Back Pain - A Double Blind, Randomised, Placebo Controlled Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E0646-AS91-301
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Muscle Spasm; Back Pain
Keywords: Muscle; Spasm; Back; Pain
MeSH Terms: conditions — Spasm; Back Pain; Pain | interventions — eperisone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Eperisone

SUMMARY:
The purpose of this study is to evaluate the efficacy of Eperisone HCl in the treatment of Acute Musculoskeletal spasm associated with Low-Back Pain.

DETAILED DESCRIPTION:
This is a multi-center trial, which will be conducted in a total of 240 patients (120 patients in each treatment group). Patients attending the out-patient setting of traumatology and orthopedic departments of the study centers will be screened for lumbar pain and spasm by clinical and radiological examination for inclusion. In this study, it has been planned to enroll a total of 240 patients with 120 patients in each group. The total duration of treatment will be 14 days. Patients will be screened for baseline parameters and will then be randomized, as per the predetermined randomization schedule, into two groups. Patients will be treated with either Eperisone-HCl (Myonal) or placebo for a period of 14 days. After the baseline-screening visit (Day 1), the patients would be asked to follow up on day 3, day 7, and day 14. During each visit, a complete general examination and clinical evaluation of efficacy parameters would be done. Adverse events would be monitored during the study period and would be recorded in the Case Report Form (CRF). At the end of the treatment, Global Assessment of Response to Therapy by Physicians and Patients (PGART) would be done for efficacy and tolerability separately.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex between 18 to 60 years of age.
2. Patients with confirmed diagnosis of Acute Musculoskeletal spasm with Low Back Pain due to:

   * Spondylosis deformans
   * Prolapsed Intervertebral Disc (PID)
   * Muscle sprains with spasms
3. Patients who are willing to take the medications as directed and willing to come for follow-ups.
4. Patients who are willing to comply with the protocol requirements.
5. Patients who are willing to give the written informed consent.

Exclusion Criteria:

1. Patients with other associated spasm conditions like:

   * Muscle sprains with spasms of hip/knee/ankle
   * Traumatic pain with spasms
   * Cervical Spondylitis
   * Pain & spasm associated with fractured bone.
2. Patients who had taken any form of skeletal muscle relaxant in the previous 7 days.
3. Patients with hypersensitivity to any of the ingredients of the test & control formulations.
4. Pregnant/Lactating women or women of child bearing potential not following adequate contraceptive measures.
5. Patients unwilling or unable to comply with the study procedures.
6. Patients having a history of severe acute infection, major surgery or trauma, severe metabolic, endocrine or electrolyte disturbances and seizures in preceding 8 weeks.
7. Patients having severe renal insufficiency defined by a creatinine value above 2.5 mg/dl.
8. Patients having severe hepatic insufficiency defined by an SGOT or SGPT value equal or higher than the threefold normal values of the respective laboratory reference value.
9. Patients having any of the following disorders:

   * Renal failure
   * Bulimia
   * Hypo and Hyperthyroidism
   * Nephrotic syndrome
   * Anorexia nervosa
   * Biliary obstruction
   * Severe cardiac dysfunction.
10. Patients having uncontrolled diabetes mellitus, or any other metabolic or endocrine disorder.
11. Patients that have received treatment with any investigational drug in the preceding 4 weeks.
12. Patients likely to be non-compliant (alcohol, smoking or drug abusers).
13. Any condition that, in the opinion of the investigator, does not justify patient's inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2006-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The present study will be conducted with an objective of comparing the efficacy of Eperisone-HCl (Myonal) versus placebo in the treatment of acute musculoskeletal spasm associated with low back pain.

SECONDARY OUTCOMES:
The present study will be conducted with a secondary objective of comparing the tolerability of Eperisone-HCl (Myonal) versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dilip Pawar, Study Director — Eisai Pharmaceuticals India Pvt. Ltd
Locations (4):
- India (4):
  - M.R. Medical College, Kalaburagi, Karnataka
  - Grant Medical College Sir J.J. Group of Hospitals, Byculla, Mumbai, Maharashtra
  - L.T. M. Medical College and General Hospital, Sion, Mumbai, Maharashtra
  - Post Graduate Institute of Medical Education and Research (PGI), Chandigarh, Punjab